CLINICAL TRIAL: NCT04291950
Title: Epigenetics of Triple-Negative Breast Cancer in Overweight and Obese Hispanic and Non-Hispanic White Women
Brief Title: Epigenetics of TNBC in Overweight and Obese Hispanic & Non-Hispanic White Women
Status: Withdrawn | Type: Observational
Why Stopped: Principal investigator is moving to a new institution. Study is closing.
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: 2001272738; 32097 (Other: University of Arizona Cancer Center)
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Triple Negative Breast Cancer
Keywords: triple negative; breast cancer; TNBC; obesity; overweight; Hispanic; non-Hispanic white
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Obesity; Overweight | interventions — Biopsy, Needle; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Four (4) 16-gauge core needle biopsies of breast tissue.
  Ten (10) ml of blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Hispanic and NHW women undergoing either a benign breast surgery or prophylactic mastectomy.
  Interventions: Procedure: Needle core biopsy
- Newly diagnosed TNBC: Hispanic and NHW with newly diagnosed TNBC. Patients with TNBC will be eligible regardless of whether their treatment plan is surgery first or chemotherapy first (neoadjuvant chemotherapy).
  Interventions: Procedure: Needle core biopsy

INTERVENTIONS:
Procedure: Needle core biopsy — Blood draws will be done in OR by research staff. Tissue will be obtained at the time of their definitive surgery or at the time of port placement. For women going to surgery first, four (4) 16-gauge core needle biopsies will be obtained by research staff after the tumor has been removed from the patient and the specimen is on the collection table in the OR.
  For women who are getting neo-adjuvant therapy prior to surgery, the core needle biopsies will be collected at the time of port placement in the OR. The patient will be under light anesthesia for the port placement. Per standard care, we will also use local anesthetic for the needle core biopsy. Port placement requires ultrasound (US). We will take advantage of the US already available in the OR to guide the core needle biopsy. Within 30 minutes of procurement, the tissue from the biopsies will be flash frozen in liquid nitrogen by staff and taken to the lab.
  Other Names: Blood draw

SUMMARY:
A key tenet of this project is that of reaching translational human diagnosis and biomarker end points. To lay a foundation and make progress towards these translational goals, investigators will address the following specific aim:

To determine if BMI/ obesity differentially influence expression and epigenetic signatures in triple negative breast cancer (TNBC) from Hispanic compared to NHW women.

DETAILED DESCRIPTION:
The intended goal of this Project is to develop epigenetic biomarkers to monitor the role of obesity and ethnicity on he development of triple negative breast cancer (TNBC). The proposed approach will seek to clarify for the first time if BMI is a biological factor that regulates aromatic hydrocarbon receptor (AhR) expression and epigenetic activity at breast cancer susceptibility and hormone receptor genes based on Hispanic or non-Hispanic white (NHW) ethnicity. If successful, the proposed experiments have the potential to highlight the role of overweight and obesity for dietary prevention of TNBC and to underscore the consideration of breast cancer screening among overweight/obese Hispanic women. Additionally, this study will provide the opportunity to begin testing the utility of AhR as a biomarker of TNBC development related to BMI and ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic or NHW women
* ≥ 18 years of age
* scheduled for a breast procedure as standard of care treatment - benign breast surgery or prophylactic mastectomy\
* Newly diagnosed TNBC - Patients with TNBC will be eligible regardless of whether their treatment plan is surgery first or chemotherapy first (neoadjuvant chemotherapy)
* Eligible non-white women could be included

Exclusion Criteria:

* BRCA1/2 mutation carriers
* Family history of breast cancer in a first-degree relative and have NOT had genetic testing for BRCA1/2
* Patients who have already undergone radiation or chemotherapy
* Pregnant women
* Male
* Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: he overall strategy for this pilot project is to collect breast tissue from 30 non-tumor (control) subjects and 30 TNBC patients. The women will be stratified by BMI (lean, overweight, obese) and ethnicity (Hispanic vs NHW). Race and ethnicity will be self-reported. Hispanic women can be of any race. Due to the Southwestern location of the University of Arizona (UA) and the regional demographics, we expect that approximately 90% of the Hispanic women recruited for this study will be White of Mexican/Mexican-American ancestry. However, eligible non-White, Hispanic or non-Hispanic, subjects will not be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08-30 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
To determine if BMI/ obesity differentially influence expression and epigenetic signatures in TNBC from Hispanic compared to NHW women. | Two years
  DXA studies will be completed prior to surgery or port placement. Blood draws will be done in OR by research staff. Tissue will be obtained at the time of their definitive surgery or at the time of port placement. For women going to surgery first, four (4) 16-gauge core needle biopsies will be obtained by research staff after the tumor has been removed from the patient and the specimen is on the collection table in the OR.
  For women who are getting neo-adjuvant therapy prior to surgery, the core needle biopsies will be collected at the time of port placement in the OR.

CONTACTS AND LOCATIONS:
Overall Officials: Pavani Chalasani, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided